CLINICAL TRIAL: NCT01545440
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of Lebrikizumab in Patients With Uncontrolled Asthma Who Are on Inhaled Corticosteroids and A Second Controller Medication
Brief Title: A Study of Lebrikizumab in Patients Whose Asthma is Uncontrolled With Inhaled Corticosteroids and A Second Controller Medication (LUTE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GB27862; 2011-004218-41 (EudraCT Number)
Record Dates: First submitted 2012-03-01; First posted 2012-03-06 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — lebrikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- lebrikizumab - highest dose (Experimental)
  Interventions: Drug: lebrikizumab
- lebrikizumab - lowest dose (Experimental)
  Interventions: Drug: lebrikizumab
- lebrikizumab - middle dose (Experimental)
  Interventions: Drug: lebrikizumab
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: lebrikizumab — subcutaneous dose every 4 weeks
  Arms: lebrikizumab - middle dose
Drug: lebrikizumab — subcutaneous dose every 4 weeks
  Arms: lebrikizumab - lowest dose
Drug: lebrikizumab — subcutaneous dose every 4 weeks
  Arms: lebrikizumab - highest dose
Drug: placebo — subcutaneous dose every 4 weeks
  Arms: placebo

SUMMARY:
This randomized, multicenter, double-blind, placebo-controlled, parallel-group study will assess the efficacy and safety of lebrikizumab in patients with asthma whose disease remains uncontrolled despite daily therapy with an inhaled corticosteroid and a second controller medication. Patients will be randomized in a 1:1:1:1 ratio to receive double-blind treatment with subcutaneous lebrikizumab ("highest", "middle", "lowest" dose) or placebo every 4 weeks for 52 weeks, in addition to their standard-of-care therapy. This will be followed by a 52-week double-blind active treatment extension. The anticipated time on study treatment is up to 104 weeks. There will be a safety follow-up of 24 weeks after the last dose of study drug for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 to 75 years of age at Visit 1
* Asthma diagnosis for >/= 12 months prior to the start of screening (Visit 1)
* Bronchodilator response during screening
* Pre-bronchodilator FEV1 40%-80% of predicted during screening
* On ICS (inhaled corticosteroids) 500-2000 mcg/day of fluticasone propionate DPI or equivalent for >/= 6 months prior to the start of screening (Visit 1) with no anticipated changes throughout the study
* On an eligible second controller medication (LABA, LAMA, LTRA or theophylline within the prescribed dosing range)
* Uncontrolled asthma as defined by protocol both during screening period and at time of randomization
* Chest X-ray or computed tomography (CT) scan obtained within 12 months prior to screening or chest X-ray during screening period confirming the absence of other lung disease
* Demonstrated adherence with controller medication during the screening period

Exclusion Criteria:

* History of severe allergic or anaphylactic reaction to a biologic agent or known hypersensitivity to any component of the lebrikizumab injection
* Use of zileuton or roflumilast within 6 months prior to screening
* Maintenance oral corticosteroid therapy, defined as daily or alternate day oral corticosteroid maintenance therapy within the 3 months prior to Visit 1
* Treatment with systemic (oral, intravenous or intramuscular) corticosteroids within the 4 weeks prior to Visit 1
* Major episode of infection within 4 weeks prior to Visit 1 or treatment with oral antibiotics within 2 weeks prior to Visit 1
* Active parasitic infection within the 6 months prior to Visit 1
* Active tuberculosis requiring treatment within the 12 months prior to Visit 1
* Known immunodeficiency, including, but not limited to, HIV infection
* Evidence of acute or chronic hepatitis or known liver cirrhosis
* History of cystic fibrosis, chronic obstructive pulmonary disease, and/or other clinically significant lung disease other than asthma
* Known malignancy or current evaluation for a potential malignancy
* Current smoker or former smoker with a history >10 pack years
* History of alcohol, drug or chemical abuse
* Initiation or change in allergen immunotherapy within 3 months prior to Visit 1
* Use of biologic therapy including omalizumab during 6 months prior to Visit 1
* Receipt of live/attenuated vaccine within 4 weeks prior to Visit 1
* Pregnant or lactating women
* Body mass index (BMI) > 38 kg/m2
* Body weight < 40 kg

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Rate of asthma exacerbations during the 52-week placebo-controlled period | weeks 0-52

SECONDARY OUTCOMES:
Change in lung function: pre-bronchodilator FEV1 | from baseline to week 52
Time to first asthma exacerbation | from baseline to week 52
Change in fractional exhaled nitric oxide (FeNO) | from baseline to week 52
Change in asthma-specific health-related quality of life, assessed by the Standardized Asthma Quality of Life Questionnaire (AQLQ[S]) | from baseline to week 52
Change in asthma rescue medication use | from baseline to week 52
Rate of urgent asthma-related health care utilization during the 52-week placebo-controlled period | from baseline to week 52

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (67):
- United States (66):
  - Pell City, Alabama
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Bakersfield, California
  - Fountain Valley, California
  - Fullerton, California
  - Los Angeles, California
  - Mission Viejo, California
  - Napa, California
  - Orange, California
  - Rancho Mirage, California
  - Sacramento, California
  - San Diego, California
  - Studio City, California
  - Upland, California
  - Walnut Creek, California
  - Centennial, Colorado
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Wheat Ridge, Colorado
  - Waterbury, Connecticut
  - Gainesville, Florida
  - North Palm Beach, Florida
  - Ocala, Florida
  - Tallahassee, Florida
  - Tampa, Florida
  - Winter Park, Florida
  - Albany, Georgia
  - Savannah, Georgia
  - Honolulu, Hawaii
  - River Forest, Illinois
  - Topeka, Kansas
  - Metairie, Louisiana
  - Bangor, Maine
  - Kansas City, Missouri
  - Bellevue, Nebraska
  - Las Vegas, Nevada
  - Albuquerque, New Mexico
  - Great Neck, New York
  - New York, New York
  - Rockville Centre, New York
  - The Bronx, New York
  - High Point, North Carolina
  - Wilmington, North Carolina
  - Cincinnati, Ohio
  - Eugene, Oregon
  - Lake Oswego, Oregon
  - Portland, Oregon
  - Blue Bell, Pennsylvania
  - Easton, Pennsylvania
  - Harrisburg, Pennsylvania
  - Philadelphia, Pennsylvania
  - Upland, Pennsylvania
  - Warwick, Rhode Island
  - Greenville, South Carolina
  - Spartanburg, South Carolina
  - Knoxville, Tennessee
  - Arlington, Texas
  - Dallas, Texas
  - El Paso, Texas
  - Fort Worth, Texas
  - McKinney, Texas
  - San Antonio, Texas
  - Henrico, Virginia
  - Seattle, Washington
  - Madison, Wisconsin
- Nedlands, Western Australia, Australia

REFERENCES:
- [Derived] Chen M, Shepard K 2nd, Yang M, Raut P, Pazwash H, Holweg CTJ, Choo E. Overlap of allergic, eosinophilic and type 2 inflammatory subtypes in moderate-to-severe asthma. Clin Exp Allergy. 2021 Apr;51(4):546-555. doi: 10.1111/cea.13790. Epub 2021 Jan 7. PMID 33217063
- [Derived] Hanania NA, Noonan M, Corren J, Korenblat P, Zheng Y, Fischer SK, Cheu M, Putnam WS, Murray E, Scheerens H, Holweg CT, Maciuca R, Gray S, Doyle R, McClintock D, Olsson J, Matthews JG, Yen K. Lebrikizumab in moderate-to-severe asthma: pooled data from two randomised placebo-controlled studies. Thorax. 2015 Aug;70(8):748-56. doi: 10.1136/thoraxjnl-2014-206719. Epub 2015 May 22. PMID 26001563
- See also: study website — http://myasthmastudies.com